CLINICAL TRIAL: NCT01352182
Title: Pharmacokinetic Characteristics of Pioglitazone and Preliminary Biomarker Response in Adolescents Aged 12 to 17 Years With Severe Sepsis and Septic Shock
Brief Title: Pharmacokinetic and Biomarker Study of Pioglitazone in Adolescents With Severe Sepsis and Septic Shock
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PIOSEPSIS1217
Record Dates: First submitted 2011-02-23; First posted 2011-05-11 (Estimated); Results first posted 2020-09-02 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Severe Sepsis; Septic Shock
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pioglitazone hydrochloride (Experimental): Pioglitazone hydrochloride treatment group
  Interventions: Drug: Pioglitazone hydrochloride
- Normal standard care (No Intervention): Normal standard care control group

INTERVENTIONS:
Drug: Pioglitazone hydrochloride — Participants will receive a daily dose of pioglitazone at 0.5 mg/kg/dose for 5 days.
  Other Names: Actos
  Arms: Pioglitazone hydrochloride

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics of pioglitazone and to determine the effect on inflammatory biomarkers for pioglitazone in patients with severe sepsis and septic shock.

DETAILED DESCRIPTION:
Severe sepsis is a major cause of morbidity and mortality among adults and children. Few clinical trials have demonstrated clinical benefit in sepsis. Severe sepsis is a systemic inflammatory syndrome in response to infection that is associated with acute organ dysfunction. The nuclear receptor peroxisome proliferator-activated receptor-gamma (PPARg) is involved in the regulation of the sepsis-induced inflammatory response. The central hypothesis is that pioglitazone reduces the inflammatory responses in children with severe sepsis and septic shock.

ELIGIBILITY:
Inclusion Criteria:

* Weight range between 30 to less than or equal to 90kg
* Have a known or suspected infection and meet criteria for severe sepsis or septic shock as defined according to the International Pediatric Sepsis Consensus Conference guidelines

Exclusion Criteria:

* Are in a moribund state in which death is perceived as imminent
* Have an advanced directive or do not resuscitate order to withhold life-sustaining
* Have a history of cyanotic heart disease or congestive heart failure
* Have a serum transaminase level (ALT) that exceeds about 2.5 times the upper limit of normal (>112 unit/L)
* Are or become pregnant
* Are already on or have a history of taking pioglitazone or rosiglitazone
* Have type 1 or 2 diabetes
* Have total body weight below 30 kg or above 90 kg
* Have a serious condition, in addition to sepsis, which in the opinion of the investigator would compromise the participant

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-10; Primary Completion 2016-05 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer M. Kaplan, M.D., M.S., Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Background] Kaplan JM, Denenberg A, Monaco M, Nowell M, Wong H, Zingarelli B. Changes in peroxisome proliferator-activated receptor-gamma activity in children with septic shock. Intensive Care Med. 2010 Jan;36(1):123-30. doi: 10.1007/s00134-009-1654-6. Epub 2009 Sep 17. PMID 19760394
- [Background] Sherwin CM, Ding L, Kaplan J, Spigarelli MG, Vinks AA. Optimal study design for pioglitazone in septic pediatric patients. J Pharmacokinet Pharmacodyn. 2011 Aug;38(4):433-47. doi: 10.1007/s10928-011-9202-8. Epub 2011 Jun 11. PMID 21667139
- [Result] Kaplan JM, Zingarelli B, Krallman K, Tang Girdwood S, Lagory D, Mizuno T, Fei L, Wong HR, Vinks AA. Phase 1 safety and pharmacokinetic study on the use of pioglitazone in critically ill patients with sepsis: a randomized clinical trial. Intensive Care Med. 2018 Nov;44(11):2006-2008. doi: 10.1007/s00134-018-5374-7. Epub 2018 Sep 25. No abstract available. PMID 30255316
- See also: Kaplan Lab Page — http://www.cincinnatichildrens.org/research/divisions/c/critical/labs/Kaplan/default/

RESULTS

PARTICIPANT FLOW:
Groups:
- Normal Standard Care: Received normal routine standard care
Period: Overall Study
Arm/Group | Pioglitazone Hydrochloride | Normal Standard Care
Started | 8 | 4
Completed | 8 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Normal Standard Care: Routine normal standard care
- Total: Total of all reporting groups
Arm/Group | Pioglitazone Hydrochloride | Normal Standard Care | Total
Number analyzed (Participants) | 8 | 4 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.8 (3.5) | 20.8 (9.7) | 16.083 (6.721)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 5 | 1 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 4 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 4 | 12

OUTCOME MEASURES:

1. Primary Outcome: Evaluate the Safety Profile of Pioglitazone in Patients With Severe Sepsis and Septic Shock as the Number of Hypoglycemic Events
Description: The number of hypoglycemic events in pioglitazone vs standard care. Hypoglycemia was defined as blood glucose level that remains <40mg/dl despite dextrose bolus treatment.
Time Frame: Assessement over five days
Population: Hypoglycemia episodes
Measure: Number; unit: events
Arm/Group | Pioglitazone Hydrochloride | Normal Standard Care
Number analyzed (Participants) | 8 | 4
events | 0 | 0
Statistical Analysis 1: Comparison: Pioglitazone Hydrochloride vs Normal Standard Care; Test type: Superiority; p = 1.0, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Safety Labs - Blood Urea Nitrogen (BUN)
Description: BUN levels in blood from subject on the final day of enrollment
Time Frame: Final day of study
Measure: Median (Inter-Quartile Range); unit: mg/dl
Arm/Group | Pioglitazone Hydrochloride | Normal Standard Care
Number analyzed (Participants) | 8 | 4
mg/dl | 7.5 [6 to 18.75] | 10 [5.25 to 15.5]
Statistical Analysis 1: Comparison: Pioglitazone Hydrochloride vs Normal Standard Care; Test type: Superiority; p = 1.0, Wilcoxon (Mann-Whitney) — threshold for significance p<0.05

3. Primary Outcome: Safety Labs - Creatinine
Description: Creatinine levels in blood from subject on the final day of enrollment
Time Frame: Final day of study
Measure: Median (Inter-Quartile Range); unit: mg/dl
Arm/Group | Pioglitazone Hydrochloride | Normal Standard Care
Number analyzed (Participants) | 8 | 4
mg/dl | 0.72 [0.39 to 0.778] | 0.415 [0.305 to 0.593]
Statistical Analysis 1: Comparison: Pioglitazone Hydrochloride vs Normal Standard Care; Test type: Superiority; p = 0.154, Wilcoxon (Mann-Whitney) — threshold for significance p<0.05

4. Primary Outcome: Safety Labs - Alanine Aminotransferase (ALT)
Description: ALT levels in blood from subject on the final day of enrollment
Time Frame: Final day of study
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | Pioglitazone Hydrochloride | Normal Standard Care
Number analyzed (Participants) | 8 | 4
U/L | 21.5 [13.5 to 25.25] | 24.5 [11 to 27.5]
Statistical Analysis 1: Comparison: Pioglitazone Hydrochloride vs Normal Standard Care; Test type: Superiority; p = 0.683, Wilcoxon (Mann-Whitney) — significance threshold p<0.05

5. Primary Outcome: Pioglitazone Area Under Curve Estimates by Treatment Group and Route of Administration
Description: Pioglitazone concentration as the total area under curve divided by the number of days receiving the drug in subjects who took the drug by mouth versus by naso-gastric tube
Time Frame: five days
Measure: Mean (Standard Deviation); unit: ng*h/ml
Groups:
- Pioglitazone Hydrochloride by Mouth: Pioglitazone hydrochloride: Participants will receive a daily dose of pioglitazone at 0.5 mg/kg/dose for 5 days taken by mouth
- Pioglitazone Hydrochloride by Nasogastric Tube: Pioglitazone hydrochloride: Participants will receive a daily dose of pioglitazone at 0.5 mg/kg/dose for 5 days taken by nasogastric tube
Arm/Group | Pioglitazone Hydrochloride by Mouth | Pioglitazone Hydrochloride by Nasogastric Tube
Number analyzed (Participants) | 5 | 3
ng*h/ml | 5363 (2362) | 1052 (942)
Statistical Analysis 1: Comparison: Pioglitazone Hydrochloride by Mouth vs Pioglitazone Hydrochloride by Nasogastric Tube; Test type: Superiority; p = 0.08, t-test, 2 sided — significance threshold p<0.05

6. Secondary Outcome: Effect of Pioglitazone Area Under the Curve on Changes in IL-6
Description: We examined the effect of pioglitazone Area under the curve on IL-6 in patients receiving pioglitazone only. (Control subjects did not receive pioglitazone). The pharmacokinetic endpoint was area under the curve (AUC) total/days of pioglitazone administration
Time Frame: Evaluation of inflammatory biomarkers will be obtained prior to dosing for the first five days of the study
Population: Log interleukin (IL)-6. The pharmacokinetic endpoint was area under the curve (AUC) total/days of pioglitazone administration
Measure: Least Squares Mean (Standard Error); unit: ng/ml
Arm/Group | Pioglitazone Hydrochloride | Normal Standard Care
Number analyzed (Participants) | 8 | 4
ng/ml | -1.4425 (0.3741) | NA (NA) — patient in the normal standard care group did not receive pioglitazone
Statistical Analysis 1: Comparison: Pioglitazone Hydrochloride; Test type: Other — linear regression; p = 0.003, Regression, Linear; Slope = -1.44, Standard Error of Mean 0.3741

ADVERSE EVENTS:
Time Frame: Adverse events were monitored for each subject throughout each subject's hospitalization which ranged from 4 days to 30 days for control subjects and 4 days to 23 days for pioglitazone subjects.
Arm/Group | Pioglitazone Hydrochloride | Normal Standard Care
All-Cause Mortality (participants affected / at risk) | 2/8 | 0/4
Serious Adverse Events (participants affected / at risk) | 2/8 | 0/4
Other Adverse Events (participants affected / at risk) | 5/8 | 2/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pioglitazone Hydrochloride (N=8) | Normal Standard Care (N=4)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Severe biventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
mediastinal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Surgical and medical procedures - Other (Surgical and medical procedures) | 1 (1) | 0 (0)
ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
hemolysis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
intracranial hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pioglitazone Hydrochloride (N=8) | Normal Standard Care (N=4)
Anemia (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
Complaint of chest pain (Cardiac disorders) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Edema (General disorders) | 1 (1) | 1 (1)
Fever (General disorders) | 5 (5) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
INR increased (Investigations) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 2 (2) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Weight gain (Investigations) | 1 (1) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Alkalosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Renal and urinary disorders - other, increased BUN (Renal and urinary disorders) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hpoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Mild pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Edema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - other, skin breakdown and oozing (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischemia (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Small sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No